CLINICAL TRIAL: NCT02618642
Title: The Use of i/t Curve in Assessment of Effects of Biceps Brachii Phototherapy With PILER Light
Brief Title: The Use of i/t Curve in Assessment of Phototherapy Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Jolanta Zwolińska, PhD, University of Rzeszow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: jz.i/t
Record Dates: First submitted 2015-11-27; First posted 2015-12-01 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Nerve Disorders
Keywords: electrodiagnostics; i/t curve; neuromuscular excitation; PILER (Polychromatic Incoherent Low-Energy Radiation); algometry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A total of the 120 participants who agreed to fulfil the inclusion criteria throughout the study were randomly chosen by drawing marked squares from an opaque envelope. They were helped by an assistant researcher. The sixty individuals were selected in this way Next, those who were enrolled were further randomized into four groups, each including 15 individuals:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Piler light + red filter (Active Comparator): Group x: irradiation with a red filter (visible red radiation and infrared; 650-800 nm and 800-3900 nm, respectively) time of phototherapy treatment: 10 minutes for one session 10 irradiations to the biceps brachii muscle
  Interventions: Radiation: Irradiations of the biceps brachii muscle with PILER light. The participants were randomized into 4 groups: group v - no filter/ group x - red filter/ group y - blue filter/ group z - placebo.
- Piler light + blue filter (Active Comparator): Group y: irradiation with a blue filter (blue radiation; 440-480 nm) time of phototherapy treatment: 10 minutes for one session 10 irradiations to the biceps brachii muscle
  Interventions: Radiation: Irradiations of the biceps brachii muscle with PILER light. The participants were randomized into 4 groups: group v - no filter/ group x - red filter/ group y - blue filter/ group z - placebo.
- Piler light without a filter (Active Comparator): Group v: irradiation without a filter (white radiation in the entire spectrum and near-infrared radiation; 480-3400 nm) one session lasted 10 minutes 10 irradiations to the biceps brachii muscle
  Interventions: Radiation: Irradiations of the biceps brachii muscle with PILER light. The participants were randomized into 4 groups: group v - no filter/ group x - red filter/ group y - blue filter/ group z - placebo.
- placebo (Placebo Comparator): Group z: placebo irradiation (without a filter, 3 min, distance: 100 cm). time of phototherapy treatment: 3 minutes for one session distance of 1meter 10 irradiations to the biceps brachii muscle
  Interventions: Radiation: Irradiations of the biceps brachii muscle with PILER light. The participants were randomized into 4 groups: group v - no filter/ group x - red filter/ group y - blue filter/ group z - placebo.

INTERVENTIONS:
Radiation: Irradiations of the biceps brachii muscle with PILER light. The participants were randomized into 4 groups: group v - no filter/ group x - red filter/ group y - blue filter/ group z - placebo. — Biceps brachii examination was carried out before (examination 1) and after (examination 2) a series of 10 PILER light treatments. It included a traditional electrodiagnostic examination and the assessment of the pressure pain threshold (PPT).
  The electrodiagnostic examination of the muscle was performed using the unipolar stimulation method from the direct motor point. The passive electrode (6 cm x 6 cm) was attached to the side of the distal part of the forearm, and the distal edge of the electrode was adjacent to the proximal edge of the ulnar styloid process. The examination was performed with a Multitronic MT3 electrotherapy apparatus set.
  PPT at the direct motor point was determined using an algometer (Algometer commander TM ITECH Medical Industries). A head with a rubber jacket with a surface area of 0.5 cm2 was used to cause pressure pain. Pressure was exerted until the participant reported pain, at which time the force (lbs) marked by the algometer was recorded.

SUMMARY:
Conventional electrodiagnostic examination is useful in daily physiotherapeutic practice. Nevertheless, the subjective assessment of muscle contraction and perceived current vibrations carries the risk of error and thus is a limitation of the method. Therefore, the use of the I/T curve coefficient was proposed in this study. This coefficient is the arithmetic mean of the electrical charge needed to trigger a sensory or motor reaction at different widths of the electrical pulse. PILER (Polychromatic Incoherent Low-Energy Radiation) light affects the sensory and motor excitability of the tissue. The resulting changes may depend on the colour of the filter used in the irradiations.

The study aimed to:

1. To evaluate changes in neuromuscular excitability occurring after PILER irradiation using filters of different colours.
2. To evaluate the usefulness of the I/T curve coefficient in neuromuscular excitation test.

60 healthy volunteers were assigned to one of four groups irradiated with: 1 - Piler light + red filter, 2 - Piler light + blue filter, 3 - Piler light without a filter, 4 - placebo.

Main Outcome Measures were plotting I/T curve coefficient for rectangular (■I/T coeff) and triangular (▲I/T coeff) pulses and the pressure pain threshold (PPT).

DETAILED DESCRIPTION:
Electrodiagnostic examination is a valuable addition to clinical trials and is useful in disorders of neuromuscular excitability.

The I/T curve is a non-invasive electrodiagnostic method for the quantitative assessment of neuromuscular excitation. Plotting it makes it possible to determine the rheobase (minimum stimulus amplitude to reach the stimulation threshold with a long pulse duration /1000 ms/) and chronaxie (minimum duration of a stimulus with an amplitude twice that of the rheobase needed to reach the stimulation threshold.

Traditional electrodiagnostic examination is popular among clinicians due to its availability, ease of administration and usefulness in physiotherapeutic practice. The subjective assessment of muscle contraction and perceived current vibrations carries the risk of error and thus is a limitation of the method. Therefore, use of the I/T curve coefficient was proposed in this study. This coefficient is the arithmetic mean of the electrical charge needed to trigger a sensory or motor reaction at different widths of the electrical pulse.

Polarized polychromatic incoherent low-energy radiation (PILER light) can affect the sensory and motor excitability of living tissue. The biological activity of light results from the energy of its ordered electromagnetic waves acting on living cells. No thermal effect is present, as the density of the energy transmitted to the tissues is low.PILER therapy often uses filters of different colours, each showing a slightly different effect on excitable tissue.

The research questions of this randomised experiment were:

1. Does PILER light affect sensory and motor excitation?
2. Does the electromagnetic wavelength of PILER light influence its effect?
3. Is the I/T curve coefficient a useful measure of sensory and motor excitation?

ELIGIBILITY:
Inclusion Criteria included: informed consent, good tolerance of current pulses, completion of all phototherapy sessions, declaration of alcohol/drugs/smoking abstinence

The exclusion criteria were: acute inflammatory processes and fever, the presence of pigmented moles in the irradiated area, exposure to any other physical factors, a history of upper limb trauma, and upper limb overload.

Ages: 21 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 participants meeting inclusion criteria (healthy volunteers) were randomized into 4 groups
  Setting: Centre for Innovative Research in Medical and Natural Sciences, the University of Rzeszów Faculty of Medicine, Poland.
Groups:
- PILER Light Irradiation Treatments With Red Filter: Group x: Participants received a series of 10 PILER light (polychromatic incoherent low-energy radiation) irradiation with a red filter (visible red radiation and infrared; 650-800 nm and 800-3900 nm, respectively), each session lasted 10 minutes,
- PILER Light Irradiation Treatments With Blue Filter: Group y: Participants received a series of 10 PILER light (polychromatic incoherent low-energy radiation) irradiation with a blue filter (blue radiation; 440-480 nm), each session lasted 10 minutes,
- PILER Light Irradiation Treatments Without a Filter: Group v: Participants received a series of 10 PILER light (polychromatic incoherent low-energy radiation) irradiation without filter (white radiation in the entire spectrum and near-infrared radiation; 480-3400 nm), each session lasted 10 minutes,
- Placebo: Group z: placebo irradiation (without a filter, 3 min, distance: 100 cm); each session lasted 3 minutes
Period: Before 10 PILER Irradiation Treatments
Arm/Group | PILER Light Irradiation Treatments With Red Filter | PILER Light Irradiation Treatments With Blue Filter | PILER Light Irradiation Treatments Without a Filter | Placebo
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0
Period: After 10 PILER Irradiation Treatments
Arm/Group | PILER Light Irradiation Treatments With Red Filter | PILER Light Irradiation Treatments With Blue Filter | PILER Light Irradiation Treatments Without a Filter | Placebo
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group x: PILER Irradiation Treatments With Red Filter: Piler light + red filter Group x: irradiation with a red filter (visible red radiation and infrared; 650-800 nm and 800-3900 nm, respectively) time of phototherapy treatment: 10 minutes for one session 10 irradiations to the biceps brachii muscle
- Group y: PILER Irradiation Treatments With Blue Filter: Piler light + blue filter Group y: irradiation with a blue filter (blue radiation; 440-480 nm) time of phototherapy treatment: 10 minutes for one session 10 irradiations to the biceps brachii muscle
- Group v: PILER Irradiation Treatments Without a Filter: Piler light without a filter Group v: irradiation without a filter (white radiation in the entire spectrum and near-infrared radiation; 480-3400 nm) one session lasted 10 minutes 10 irradiations to the biceps brachii muscle
- Group z: Placebo: placebo Group z: placebo irradiation (without a filter, 3 min, distance: 100 cm). time of phototherapy treatment: 3 minutes for one session distance of 1meter 10 irradiations to the biceps brachii muscle
- Total: Total of all reporting groups
Arm/Group | Group x: PILER Irradiation Treatments With Red Filter | Group y: PILER Irradiation Treatments With Blue Filter | Group v: PILER Irradiation Treatments Without a Filter | Group z: Placebo | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 15 | 15 | 60
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 22 [22 to 22] | 22.5 [22 to 23] | 22 [21 to 23] | 22 [21 to 23] | 22 [21 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 11 | 11 | 41
  Male | 5 | 6 | 4 | 4 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Poland | 15 | 15 | 15 | 15 | 15
sensory i/t curve coefficient for rectangle [Mean (Standard Deviation); unit: Coulomb] — Based on the results of the electrodiagnostic test, an I/T curve was plotted for rectangular (■) pulses.The I/T curve coefficient was calculated as the mean value of the electric charge that caused the sensory response (notification by the subject of the sensation of current vibrations), according to the following equations:
  ■I/T coeff = (q1+q2 +…+q13 )/13 where pulse current × pulse duration = q in coulombs
  Coulomb | 0.0005 (0.0002) | 0.0006 (0.0002) | 0.0006 (0.0005) | 0.0005 (0.0003) | 0.0005 (0.0003)
sensory i/t curve coefficient for triangle [Mean (Standard Deviation); unit: Coulomb] — Measure Description: Measure Description: Based on the results of the electrodiagnostic test, an I/T curve was plotted for rectangular (▲) pulses.The I/T curve coefficient was calculated as the mean value of the electric charge that caused the sensory response (notification by the subject of the sensation of current vibrations), according to the following equations:
  ▲I/T coeff = (q1+q2 +…+q13 )/13 where pulse current × pulse duration = q in coulombs
  Coulomb | 0.0012 (0.0007) | 0.0010 (0.0004) | 0.0015 (0.0014) | 0.0012 (0.0008) | 0.0012 (0.0009)
motor i/t curve coefficient for rectangle [Mean (Standard Deviation); unit: Coulomb] — Measure Description: Based on the results of the electrodiagnostic test, an I/T curve was plotted for rectangular (■) pulses.The I/T curve coefficient was calculated as the mean value of the electric charge that caused the motor response (threshold muscle contraction), according to the following equations:
  ■I/T coeff = (q1+q2 +…+q13 )/13 where pulse current × pulse duration = q in coulombs
  Coulomb | 0.0009 (0.0003) | 0.00013 (0.0004) | 0.0005 (0.0002) | 0.0009 (0.0003) | 0.0009 (0.0004)
motor i/t curve coefficient for triangle [Mean (Standard Deviation); unit: Coulomb] — Measure Description: Measure Description: Based on the results of the electrodiagnostic test, an I/T curve was plotted for rectangular (▲) pulses.The I/T curve coefficient was calculated as the mean value of the electric charge that caused the motor response (threshold muscle contraction), according to the following equations:
  ▲I/T coeff = (q1+q2 +…+q13 )/13 where pulse current × pulse duration = q in coulombs
  Coulomb | 0.0034 (0.0012) | 0.0035 (0.0015) | 0.0021 (0.0007) | 0.0035 (0.0015) | 0.0031 (0.0013)
Sensory Pain Pressure Threshold [Mean (Standard Deviation); unit: lbs] | 7.2 (2.8) | 8.3 (3.2) | 9.8 (3.6) | 9.9 (5.2) | 8.8 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Pressure Pain Threshold (PPT)
Description: Increase in PPT meant decrease in sensitivity to pressure in the muscle. Decrease in PPT meant increase in sensitivity to pressure in the muscle.
Time Frame: baseline measurement and 3 weeks after a series of 10 phototherapy treatments
Measure: Mean (Standard Deviation); unit: lbs
Groups:
- Piler Light + Red Filter: Radiation: Piler light phototherapy Piler light (polychromatic incoherent low-energy radiation) + red filter time of phototherapy treatment: 10 minutes for one session
  Piler light phototherapy: Piler light + red filter: phototherapy, 10 treatment sessions,10 minutes for one session Piler light + blue filter: phototherapy, 10 treatment sessions,10 minutes for one session Piler light without a filter: phototherapy, 10 treatment sessions, 10 minutes for one session
  Piler light + red filter: 10 people Piler light + blue filter: 10 people Piler light without a filter: 10 people
- Piler Light + Blue Filter: Radiation: Piler light phototherapy Piler light (polychromatic incoherent low-energy radiation)+ blue filter time of phototherapy treatment: 10 minutes for one session
  Piler light phototherapy: Piler light + red filter: phototherapy, 10 treatment sessions,10 minutes for one session Piler light + blue filter: phototherapy, 10 treatment sessions,10 minutes for one session Piler light without a filter: phototherapy, 10 treatment sessions, 10 minutes for one session
  Piler light + red filter: 10 people Piler light + blue filter: 10 people Piler light without a filter: 10 people
- Piler Light Without a Filter: Radiation: Piler light phototherapy Piler light (polychromatic incoherent low-energy radiation)without a filter time of phototherapy treatment: 10 minutes for one session
  Piler light phototherapy: Piler light + red filter: phototherapy, 10 treatment sessions,10 minutes for one session Piler light + blue filter: phototherapy, 10 treatment sessions,10 minutes for one session Piler light without a filter: phototherapy, 10 treatment sessions, 10 minutes for one session
  Piler light + red filter: 10 people Piler light + blue filter: 10 people Piler light without a filter: 10 people
- Placebo: 3 min irradiation with Piler light from 1 meter
Arm/Group | Piler Light + Red Filter | Piler Light + Blue Filter | Piler Light Without a Filter | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
lbs | 0.0 (2.0) | -0.5 (1.6) | -1.3 (3.7) | -0.6 (2.6)
Statistical Analysis 1: Comparison: Piler Light + Red Filter vs Piler Light + Blue Filter vs Piler Light Without a Filter vs Placebo; the results in the irradiated group (n=45) and the control group (n=15) were compared; Test type: Superiority; p = 0.3879, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Piler Light + Red Filter vs Piler Light + Blue Filter vs Piler Light Without a Filter; comparison was conducted of the results obtained with a different filter were compared; Test type: Superiority; p = 0.5361, Kruskal-Wallis

2. Primary Outcome: Calculation of Sensory i/t Curve Coefficient for Rectangle (■I/T Coeff)
Description: Based on the results of the electrodiagnostic test, sensory I/T curve was plotted for rectangular (■) pulses.The I/T curve coefficient was calculated as the mean value of the electric charge that caused the sensory response (notification by the subject of the sensation of current vibrations) according to the following equations:■I/T coeff = (q1+q2 +…+q13 )/13 , where pulse current × pulse duration = q in coulombs. Comparisons were made based on the changes in the ■I/T coeff, observed as a result of PILER irradiations.
Time Frame: baseline measurement and 3 weeks after a series of 10 phototherapy treatments
Measure: Mean (Standard Deviation); unit: Coulomb
Groups:
- PILER Light Irradiation Treatments With Red Filter: Piler light + red filter Radiation: Piler light phototherapy Piler light (polychromatic incoherent low-energy radiation) + red filter time of phototherapy treatment: 10 minutes for one session
- PILER Light Irradiation Treatments With Blue Filter: Piler light + blue filter Radiation: Piler light phototherapy Piler light (polychromatic incoherent low-energy radiation)+ blue filter time of phototherapy treatment: 10 minutes for one session
- PILER Light Irradiation Treatments Without a Filter: Piler light without a filter Radiation: Piler light phototherapy Piler light (polychromatic incoherent low-energy radiation)without a filter time of phototherapy treatment: 10 minutes for one session
Arm/Group | PILER Light Irradiation Treatments With Red Filter | PILER Light Irradiation Treatments With Blue Filter | PILER Light Irradiation Treatments Without a Filter | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Coulomb | 0.0007 (0.0004) | 0.0008 (0.0002) | 0.0006 (0.0003) | 0.0001 (0.0004)
Statistical Analysis 1: Comparison: PILER Light Irradiation Treatments With Red Filter vs PILER Light Irradiation Treatments With Blue Filter vs PILER Light Irradiation Treatments Without a Filter vs Placebo; the results in the irradiated group (n=45) vs the control group (placebo) (n=15) were compared; Test type: Superiority; p = 0.4669, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: PILER Light Irradiation Treatments With Red Filter vs PILER Light Irradiation Treatments With Blue Filter vs PILER Light Irradiation Treatments Without a Filter; Test type: Superiority; p = 0.4161, Kruskal-Wallis

3. Primary Outcome: Calculation of Sensory I/T Curve Coefficient for Triangular (▲I/T Coeff) Pulses
Description: Based on the results of the electrodiagnostic test, sensory I/T curve was plotted for triangular (▲I/T coeff) pulses.The I/T curve coefficient was calculated as the mean value of the electric charge that caused the sensory response (notification by the subject of the sensation of current vibrations) according to the following equations:▲I/T coeff = (q1+q2+… +q10) /10 , where pulse current × pulse duration = q in coulombs. Comparisons were made based on the changes in the ▲I/T coeff, observed as a result of PILER irradiations.
Time Frame: baseline measurement and 3 weeks after a series of 10 phototherapy treatments
Measure: Mean (Standard Deviation); unit: Coulomb
Arm/Group | Group x: PILER Irradiation Treatments With Red Filter | Group y: PILER Irradiation Treatments With Blue Filter | Group v: PILER Irradiation Treatments Without a Filter | Group z: Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Coulomb | 0.0014 (0.0014) | 0.0018 (0.0007) | 0.0015 (0.0007) | 0.0018 (0.0019)
Statistical Analysis 1: Comparison: Group x: PILER Irradiation Treatments With Red Filter vs Group y: PILER Irradiation Treatments With Blue Filter vs Group v: PILER Irradiation Treatments Without a Filter vs Group z: Placebo; the results in the irradiated group (n=45) and the control group (n=15) were compared; Test type: Superiority; p = 0.9596, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group x: PILER Irradiation Treatments With Red Filter vs Group y: PILER Irradiation Treatments With Blue Filter vs Group v: PILER Irradiation Treatments Without a Filter; Test type: Superiority; p = 0.0907, Kruskal-Wallis

4. Primary Outcome: Calculation of Motor i/t Curve Coefficient for Rectangle (■I/T Coeff)
Description: Based on the results of the electrodiagnostic test, motor I/T curve was plotted for rectangular (■) pulses.The I/T curve coefficient was calculated as the mean value of the electric charge that caused the motor response (threshold muscle contraction) according to the following equations:■I/T coeff = (q1+q2 +…+q13 )/13 , where pulse current × pulse duration = q in coulombs. Comparisons were made based on the changes in the ■I/T coeff, observed as a result of PILER irradiations.
Time Frame: baseline measurement and 3 weeks after a series of 10 phototherapy treatments
Measure: Mean (Standard Deviation); unit: Coulomb
Arm/Group | Group x: PILER Irradiation Treatments With Red Filter | Group y: PILER Irradiation Treatments With Blue Filter | Group v: PILER Irradiation Treatments Without a Filter | Group z: Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Coulomb | 0.0009 (0.0003) | 0.0015 (0.0003) | 0.0006 (0.0003) | 0.0007 (0.0004)
Statistical Analysis 1: Comparison: Group x: PILER Irradiation Treatments With Red Filter vs Group y: PILER Irradiation Treatments With Blue Filter vs Group v: PILER Irradiation Treatments Without a Filter vs Group z: Placebo; the results in the irradiated group (n=45) and the control group (n=15) were compared; Test type: Superiority; p = 0.0110, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group x: PILER Irradiation Treatments With Red Filter vs Group y: PILER Irradiation Treatments With Blue Filter vs Group v: PILER Irradiation Treatments Without a Filter; comparison was conducted of the results obtained with a different filter (groups v, x, y,; Test type: Superiority; p = 0.1165, Kruskal-Wallis

5. Primary Outcome: Calculation of Motor I/T Curve Coefficient for Triangular (▲I/T Coeff) Pulses
Description: Based on the results of the electrodiagnostic test, Motor I/T curve was plotted for triangular (▲I/T coeff) pulses.The I/T curve coefficient was calculated as the mean value of the electric charge that caused the motor response (threshold muscle contraction) according to the following equations:▲I/T coeff = (q1+q2+… +q10) /10 , where pulse current × pulse duration = q in coulombs. Comparisons were made based on the changes in the ▲I/T coeff, observed as a result of PILER irradiations.
Time Frame: baseline measurement and 3 weeks after a series of 10 phototherapy treatments
Measure: Mean (Standard Deviation); unit: Coulomb
Arm/Group | Group x: PILER Irradiation Treatments With Red Filter | Group y: PILER Irradiation Treatments With Blue Filter | Group v: PILER Irradiation Treatments Without a Filter | Group z: Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15
Coulomb | 0.0028 (0.0009) | 0.0050 (0.0014) | 0.0024 (0.0009) | 0.0030 (0.0019)
Statistical Analysis 1: Comparison: Group x: PILER Irradiation Treatments With Red Filter vs Group y: PILER Irradiation Treatments With Blue Filter vs Group v: PILER Irradiation Treatments Without a Filter vs Group z: Placebo; he results in the irradiated group (n=45) and the control group (n=15) were compared; Test type: Superiority; p = 0.0200, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group x: PILER Irradiation Treatments With Red Filter vs Group y: PILER Irradiation Treatments With Blue Filter vs Group v: PILER Irradiation Treatments Without a Filter; Test type: Superiority — comparison was conducted of the results obtained with a different filter (groups v, x, y,; p = 0.0014, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Piler Light + Red Filter | Piler Light + Blue Filter | Piler Light Without a Filter | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT02618642/Prot_SAP_000.pdf